CLINICAL TRIAL: NCT05741541
Title: How Would the Creation of a Follow-up Methodology in Consultation Improve the Care of the Epileptic Patient?
Acronym: MAPE
Status: Completed | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A02583-40
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observationnal study is to identify the informative and educational needs of epilepsy patients to avoid interrupting the therapeutic pathway.

The main question it aims to answer are :

* Identify the patient's expectations of a nurse specializing in epilepsy in the areas of information, predictive elements of good care and adaptation to their state of health
* Identify under-addressed or misunderstood themes
* Identify patient resources and interventions already in place
* Ensuring better continuity of care
* Improve the knowledge of patients and their relatives about the management of their pathology

After a consultation with the neurologist (as part of their usual follow-up), the participants will be referred to a nurse for a semi-directive, individual interview, lasting 30 minutes and composed of open and closed questions. The announcement of the diagnosis, the quality of life or the factors contributing to the difficulties and their repercussions on a daily basis will be discussed during the interview.

ELIGIBILITY:
Inclusion Criteria:

* Adult epileptic patients, over 18 years old
* Patients with focal or generalized epilepsy
* Patients affiliated or entitled to a social security scheme
* Patients who have received informed information about the study and who have co- signed, with the investigator, a non-objection to participation in the study
* Patients whose diagnosis has been made for at least 6 months

Exclusion Criteria:

* Patients with intellectual disabilities
* Minors
* Untreated patients, in remission
* Patients without affiliation to a social security scheme
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Epileptics patients over 18 prsenting eligiblity criteria and and whose diagnosis has been made for less than 6 months and coming from for consultation in the Hôpital Nord Franche-Comté
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
Identify the informative and educational needs of epileptic patients to avoid disrupting the therapeutic course by an interview with an nurse. | At inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-Comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: No